CLINICAL TRIAL: NCT01379404
Title: Does Bio-impedance Analysis Predict Volume Overload States and Clinically Relevant Outcomes in Septic Intensive Care Unit (ICU) Patients With Acute Kidney Injury? A Prospective Observational Study
Brief Title: Bioimpedance Analysis in Septic Intensive Care Unit (ICU) Patients
Acronym: BIOVISION
Status: Completed | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Azim Gangji, principal investigator, St. Joseph's Healthcare Hamilton
Other Study IDs: StJoseph - BIOVISION
Record Dates: First submitted 2011-06-07; First posted 2011-06-23 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Sepsis
Keywords: sepsis, fluid status, BIA, CVP
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood only for chemistry.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bioelectric Impedance Analysis — Bioimpedance devices are compact, portable, easy to use, relatively inexpensive and can be used to make repeated non-invasive measurements. Bioimpedance measures the impedance to the flow of an electric current through body fluids and consists of two components, resistance and reactance. Resistance is a measure of electrical current a substance will oppose and is inversely related to tissue fluid content. Reactance is the capacitative component of impedance and indicates energy stored by cell membranes and organelles; due to this property, reactance is associated with tissue cell mass. These raw measures provide a measure of volume as determined by vector length and the RXc graph method.

SUMMARY:
Patients with severe infections initially require large amounts of fluid as part of resuscitation. Later on however, problems may arise from excess fluid such as increased time on a ventilator and kidney damage. The amount of fluid a patient has is difficult to assess. One approach is to determine the amount of fluid that is present in a large central vein. This can be done by physical examination of the jugular veins, or by placing a catheter within the vein. Unfortunately this method is unreliable and does not predict the amount of fluid a patient has.

Bioimpedance analysis (BIA), is a device that can determine the amount of fluid in the body by measuring the body's electrical properties. It is a quick and painless test that assesses volume. The primary objective of this study is to determine if BIA measurements are associated with patient important outcomes such as time on a ventilator, risk of kidney failure requiring dialysis and death. We will also determine whether BIA is a measure of fluid status in ICU patients. This study will assess feasibility in establishing a multi-centre study assessing if BIA's role in predicting adverse outcomes and thereby prognosis and fluid status. We hypothesize that shorter vector lengths will be associated with hypervolemia and less ventilator free days.

DETAILED DESCRIPTION:
Overall Objective: Persistent hypervolemia following the initial resuscitative phase in sepsis has been shown to predict morbidity and mortality. In patients with sepsis in the intensive care unit (ICU) fluid accumulation is associated with a significant increase in duration of ventilation, development of acute kidney injury (AKI) requiring dialysis and increased ICU length of stay. It is essential to be able to identify and characterize the transition from necessary fluid resuscitation to harmful fluid volume accumulation. However, current methods for assessing volume status in the ICU are imprecise. Bioelectric impedance analysis (BIA) offers a well established and easy to perform bedside technique of volume assessment. Our main objective is to prospectively determine if bio-impedance derived measures are associated with patient important outcomes including ventilator free days, AKI requiring dialysis and overall mortality in septic ICU patients. In addition, we will also assess whether BIA derived measures of volume are associated with other measures of volume status.

Hypothesis #1: Bio-impedance derived measures (phase angle, vector length) will be predict ventilator-free days by day 30 and a composite outcome of ICU patients with AKI requiring dialysis and overall mortality .

Aim #1: To assess whether a change in bio-impedance vector length (a measure of volume status) between day 3 and day 7 post- admission to the ICU predicts ventilator-free days by day 30. Secondary outcomes are mortality, AKI and length of stay in ICU.

Hypothesis #2: BIA derived volume measures (vector length and the RXc graph method) will be associated with other clinical, invasive and biochemical measures of volume status

Aim #2: To determine if BIA derived volume measures are associated with other measures of volume status including central venous pressure, N- brain natriuretic peptide (N-BNP) and physical examination findings.

Relevance: Chronic fluid overload states in ICU patients are associated with adverse clinical outcomes including prolonged ventilation, mortality, AKI and increased length of stay in the ICU. However current methods are inadequate to assess volume status accurately. This pilot observational study will determine whether implementation of bio-impedance is useful for identifying volume overload in ICU patients with sepsis. We plan to investigate whether a correlation exists between a change in vector length between days 3 and 7 post admission to the ICU and an important patient outcome of ventilator free days within the first 30 days post-enrollment. This study will assess feasibility to inform a larger multi-centre observational trial adequately powered to evaluate volume overload states as determined by bioimpedance in ICU patients with systemic inflammatory response syndrome (SIRS) and patient-important outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* high clinical suspicion for infection
* require positive pressure ventilation
* supraclavicular central line for central venous pressure measurement

Exclusion Criteria:

* Substitute decision maker unable to consent
* amputation
* pacemaker
* pregnant
* require longterm hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (>17 years) admitted to the ICU at SJHH who present with SIRS requiring positive pressure ventilation via endotracheal tube and have a clinical suspicion of infection. Consecutive sampling.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Ventilator free days | 30 days

SECONDARY OUTCOMES:
Correlation of BIA vector length with Central venous pressure, edema score, chest x-ray score, and net fluid balance | Time of enrollment (multivariate analysis at day 2 )
  To be done by multivariate analysis at day 2 vector length measurement.
Acute Kidney Injury | 60 days
Time until ICU discharge | 60 days
Mortality | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Azim Gangji, MD, MSc, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Rochwerg B, Cheung JH, Ribic CM, Lalji F, Clarke FJ, Gantareddy S, Ranganath N, Walele A, McDonald E, Meade MO, Cook DJ, Wilkieson TT, Clase CM, Margetts PJ, Gangji AS. Assessment of Postresuscitation Volume Status by Bioimpedance Analysis in Patients with Sepsis in the Intensive Care Unit: A Pilot Observational Study. Can Respir J. 2016;2016:8671742. doi: 10.1155/2016/8671742. Epub 2016 Aug 15. PMID 27597811